CLINICAL TRIAL: NCT01829529
Title: Susceptibility Changes Among Oral Microorganisms Following Single Dose Antibiotic Prophylaxis
Brief Title: Antibiotic Prophylaxis - Amoxicillin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bodil Lund (Other)
Responsible Party: Sponsor-Investigator, Bodil Lund, Assoc. professor, Dentist, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2013-000405-23
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Healthy
Keywords: Antibiotic prophylaxis
MeSH Terms: interventions — Amoxicillin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amoxicillin (Experimental): All subjects receive one dose of 2 g Amoxicillin
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin — Amoxicillin
  Other Names: Amoxicillin, Sandoz, 1 g tablet

SUMMARY:
The hypothesis of the present study is that quantitative and qualitative oral microflora alterations and changes in antibiotic susceptibility among oral commensal microflora will occur following a single dose administration of amoxicillin.

DETAILED DESCRIPTION:
A total of 33 healthy volunteers, 16 males and 17 females, will be included. Written informed consent will be obtained from all participants.

Subjects will be excluded if they have taken antibiotics within the previous three months, are pregnant, breast-feeding or allergic against penicillin.

The participants will be given a single dose of 2 g amoxicillin. Saliva samples will be collected before administration of antibiotics (day 1) and on day 2, 5, 10, 17 and 24. Un-stimulated saliva will be accumulated in a plastic container. Concentration of amoxicillin in saliva will be measured on day 1, 2 and 5. Samples will be used for the determination of antibiotic concentration. Analyses of the sensitivities to amoxicillin and some other clinically relevant antibiotic compounds will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Healthy
* Age 18-45
* Understands the study procedure and speaks Swedish and/or English

Exclusion Criteria:

* Treatment with antibiotics within the previous three months
* Pregnant
* Breast-feeding
* Allergic against penicillin
* Concomitantly participate in another medical product study
* Treatment with any kind of medication, health food preparations or probiotics

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Quantitative and qualitative changes in the oral microflora will be determined as well as changes is susceptibility to amoxicillin among these commensals. | Day 1, 2, 5, 10, 17 and 24

SECONDARY OUTCOMES:
Concentration of amoxicillin in saliva after one dose administration of amoxicillin | Day 1, 2, 5

CONTACTS AND LOCATIONS:
Overall Officials: Margareta Hultin, Dentist, Principal Investigator — Department of Dental Medicine, Karolinska Institute
Locations (1):
- Karolinska University Hospital. Department of Dental Medicine, Stockholm, Huddinge, Sweden